CLINICAL TRIAL: NCT05193136
Title: Examination of the Relationship Between Sleep Hygiene, Sarcopenia, and Cognitive Function in Patients With Chronic Obstructive Pulmonary Disease or Idiopathic Pulmonary Fibrosis
Brief Title: Sleep Hygiene, Sarcopenia, and Cognitive Function in Respiratory Disease
Status: Recruiting | Type: Observational
Sponsor: National Hospital Organization Minami Kyoto Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-32
Record Dates: First submitted 2021-12-31; First posted 2022-01-14 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Sleep Hygiene; Sarcopenia; Cognitive Function; COPD; IPF
MeSH Terms: conditions — Sleep Hygiene; Sarcopenia; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples (serum, plasma)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We aim to clarify the relationship between sleep hygiene and the onset of sarcopenia or cognitive dysfunction using sleep time, arousal, and sleep quality as indicators in COPD or IPF patients, and clarify the effects of sleep hygiene on disease progression and life prognosis.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) and idiopathic pulmonary fibrosis (IPF) have been reported to be associated with a high rate of sleep-related disorders such as insomnia, sleep-related hypoventilation, and sleep apnea syndrome.Sleep-related disorders cause symptoms such as daytime sleepiness, decreased ADL, and depression, which causes cognitive dysfunction. Both COPD and IPF have been reported to be associated with cognitive dysfunction. Recently, it has been focused on the relationship between sleep-related disorders and sarcopenia. The relationship between sleep hygiene, cognitive dysfunction, and sarcopenia in the patients with COPD or IPF is not well understood.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with COPD or IPF.

Exclusion Criteria:

* Subjects who have been hospitalized for exacerbation of respiratory failure within 1 month of study participation
* Subjects who have already been diagnosed with sarcopenia or cognitive dysfunction
* Subjects receiving long-term oxygen therapy (LTOT) or non-invasive ventilation therapy (NIV)
* Subjects with obstructive sleep apnea who are indicated for continuous positive airway pressure (CPAP)
* Subjects with severe complications such as cardiovascular disease, liver disease, renal disease, malignancy, and neurological disease.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COPD or IPF
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Relationship between sleep time at study enrollment and onset of sarcopenia during follow-up period | Two years

SECONDARY OUTCOMES:
Relationship between sleep time at study enrollment and the onset of mild cognitive impairment during follow-up period | Two years
Relationship between sleep efficiency, arousal at the time of study enrollment and the onset of sarcopenia and mild cognitive impairment during the follow-up period | Two years
Association of sleep time, sleep efficiency, arousal at the time of study enrollment and hospitalization and death due to COPD exacerbations or IPF exacerbations during follow-up period | Two years
Relationship between sleep time, sleep efficiency, arousal at the time of study enrollment and changes in grip strength, walking speed, skeletal muscle mass and cognitive function during follow-up period | Two years
Relationship between sleep time, sleep efficiency, arousal at the time of study enrollment and changes in grip strength, walking speed, skeletal muscle mass and cognitive function at the time of study enrollment | Two years
Factors associated with the onset of sarcopenia and mild cognitive impairment during follow-up period | Two years

CONTACTS AND LOCATIONS:
Locations (1):
- National Hospital Organization Minami Kyoto Hospital, Jōyō, Kyoto, Japan